CLINICAL TRIAL: NCT05867316
Title: Supplementing Brief Psychotherapy With a Mobile App
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Massachusetts General Hospital (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Evan M. Kleiman, Ph.D., Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro2022001944; R34MH113757 (NIH)
Record Dates: First submitted 2023-04-03; First posted 2023-05-19 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Suicide and Self-harm; Emotion Regulation
Keywords: suicidal ideation; suicide attempts
MeSH Terms: conditions — Suicide; Self-Injurious Behavior; Emotional Regulation; Suicidal Ideation; Suicide, Attempted

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Unified Protocol (Experimental): Unified Protocol-based treatment, with three sessions
  Interventions: Behavioral: Unified Protocol

INTERVENTIONS:
Behavioral: Unified Protocol — Unified Protocol based treatment, modified for use in brief treatment on inpatient units

SUMMARY:
Suicide is among the leading causes of death worldwide, and the risk of suicide is highest in the period immediately following discharge from inpatient psychiatric care.1Importantly, despite the enormously elevated risk during this period, nearly 50% of patients do not attend scheduled therapy after discharge. Even among those who do attend therapy, however, the skills learned in treatment may be difficult to use during the highly distressing time leading up to and during a suicide crisis. Most traditional treatments are not designed to be effective during a suicide crisis. In order to reduce the risk of suicidal thoughts and behaviors in general and specifically during the post-discharge period, interventions are needed that: (1) are easily adhered to and (2) are accessible and effective during a suicide crisis. As such, the purpose of this research study is to test an innovative, new intervention in order to develop an effective and accessible intervention for those at high risk for suicide

ELIGIBILITY:
Inclusion Criteria:

* Adult status (18+ years)
* Admission to eligible units in our partner hospital with a reason for admission having to do with suicide risk
* The ability to speak and write English fluently,
* Ownership of and consistent access to an internet-capable smartphone (e.g., an iPhone or Android phone)

Exclusion Criteria

- The presence of any factor that impairs an individual's ability to provide informed consent and comprehend and effectively participate in the study including: an inability to speak or write English fluently, the presence of gross cognitive impairment due to florid psychosis, intellectual disability, dementia, acute intoxication, or the presence of extremely agitated or violent behavior.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-09-14 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-06-06 (Actual)

PRIMARY OUTCOMES:
Suicidal thoughts | Overall changes in momentary self-reported intensity of suicidal urges (on a 11-point scale up to 4x/ day via ecological momentary assessment) from pre- to post-EMI use, across the study period, which is approximately four weeks post discharge
  Within-person changes in momentary self-reported intensity of suicidal urges (measured on a 11-point rating scale via ecological momentary assessment) from pre- to post-EMI
Self-efficacy for managing negative emotion | Beginning of study and end-of-study, approximately four weeks post discharge
  Measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) self-efficacy for managing negative emotions scale. The scale is measured with four five-point scale items, summed to a score ranging from 4 to 20 where higher scores are better.

CONTACTS AND LOCATIONS:
Overall Officials: Evan Kleiman, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Rutgers University Behavioral Healthcare, Piscataway, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share Individual participant data that underlie the results reported in this article, after de-identification (text, tables, figures, and appendices)
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Code will be shared within three months after manuscript publication.
URL: https://osf.io/6wctf/

DOCUMENTS (1):
  • Informed Consent Form (2022-12-14): https://cdn.clinicaltrials.gov/large-docs/16/NCT05867316/ICF_000.pdf